CLINICAL TRIAL: NCT03561857
Title: Essais Clinique Pour Une Endomicroscopie Robotisée Dans la redéfinition Des Stratégies d'ExérèsE (PERSÉE) appliquée à la Chirurgie de la Prostate
Brief Title: Clinical Trial for a Robotic Endomicroscopy to Better Define Resection Strategies Applied to Urology Surgery
Acronym: PERSEE II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MKT-2018-PERSEE-02; 2018-A01242-53 (Other: ANSM)
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Confocal Laser Endomicroscopy (Experimental): All included patients will undergo probe-based Confocal Laser Endomicroscopy during Robotic-Assisted Radical Prostatectomy (RARP) or Laparoscopic Radical Prostatectomy (LRP)
  Interventions: Device: Confocal Laser Endomicroscopy

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy — The study is divided in 2 parts.
  1. Ex vivo study
     * Prostate specimens will be stained using Fluorescein
     * Images/sequences of normal and abnormal prostatic tissues, and peri-prostatic tissues will be acquired.
  2. In vivo study
     * Intravenous injection of contrast agent
     * pCLE imaging every 5mm of the NVB dissection zone.
  Other Names: probe-based Confocal Laser Endomicroscopy; CelioFlex probe; Cellvizio 100 series; pCLE

SUMMARY:
This multicenter study aimed at assessing the feasibility of Probe-based Confocal Laser Endomicroscopy (pCLE) during Robotic-Assisted Radical Prostatectomy or Laparoscopic Radical Prostatectomy for intra-operative characterisation of surgical margins.

DETAILED DESCRIPTION:
Prostate cancer is one of the most diagnosed cancer in men. Several treatments are available depending on patient's clinical features. When the cancer is localised or locally advanced, one of the possible treatment is Radical Prostatectomy. A risk of that procedure is the incomplete removal of cancer tissues due to the presence of cancer cells within the resection margin. A histological analysis of the resected prostate allows to assess surgical margins. If cancer cells comes out to the edges of the removed tissue, it is called Positive Surgical Margin (PSM). Several studies showed that PSMs are more frequent in case of extra-prostatic extensions of the cancer and are correlated with biochemical recurrence.

A study conducted on 21 patients scheduled for Robotic-Assisted Radical Prostatectomy has already demonstrated the feasibility of the intra-operative observation of microscopic features of prostatic and periprostatic tissues in vivo and ex vivo with the Cellvizio® 100 Series system combined with the CelioFlex™ probe.

The main objective of the study is to assess the feasibility and safety of pCLE technology during radical prostatectomy (RP) and to assess the diagnostic performance of pCLE technology for the definition of the resection margins.

This method could be used to guide surgeons during nerve sparing surgery and provide real-time feedback for adequate dissection of NVB. As well, ex vivo characterisation of benign and cancerous glandular structures could provide an efficient and rapid method for intra-operative surgical margin assessment

The study is divided in 2 parts:

1. Ex vivo study

   An ex vivo study will be carried out on 15 firsts prostate specimens for pathologist training and generation of ex vivo pCLE images atlas.
2. In vivo study

Prior to pCLE analysis, a contrast agent (Fluorescein) will be administered:

* by intravenous injection in each prostatic pedicles before their ligation
* topically, after NVB dissection, in a spray solution through a catheter inserted in an assistant trocar or with a soaked gauze.

The Cellvizio will be used during the NVB dissection to acquire in vivo images and sequences of prostatic tissues.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Localised or locally advanced prostate cancer
* Agreement given for Radical Prostatectomy
* Not eligible or refusing an active surveillance protocol
* having given its signed informed consent

Exclusion Criteria:

* Under 18 years
* Previously treated for PCa (hormones, EBRT, focal treatments)
* Surgical history of BPH treatment
* Known allergy to Fluorescein

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
pCLE criteria | 1 year
  Definition of pCLE criteria for normal and abnormal prostate tissues

OTHER OUTCOMES:
Ease of use of the endomicroscopy device | 1 year
  The ease of use of the endomicroscopy device will be assessed using a questionnaire that the surgeon will fill at the end of each procedure
Audio/video telecommunication quality | 1 year
  The telecommunication quality will be assessed using a questionnaire that the surgeon and the anatomopathologist will fill at the end of each procedure
Number of participants with CLE imaging-related adverse events as assessed by CTCAE v5.0 | 1 year
  The device safety will measure by assessing the occurence and severity of adverse events during the study
Stability and reproducibility of images/sequences during procedures | 1 year
  The stability and reproducibility of endomicroscopy images will be assessed using a questionnaire that the surgeon and the anatomopathologist will fill at the end of each procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eric Barret, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (2):
- France (2):
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Institut Mutualiste Montsouris, Paris